CLINICAL TRIAL: NCT04251793
Title: Therapeutic Peri-implant Maintenance with Laser Therapy: an Extension of the LARST Study
Brief Title: Therapeutic Peri-implant Maintenance with Laser Therapy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Morita J USA (Unknown)
Responsible Party: Principal Investigator, Chin-Wei Wang, Clinical Assistant Professor of Dentistry, University of Michigan
Other Study IDs: HUM00160290
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2021-07

CONDITIONS: Peri-Implantitis
Keywords: Laser
MeSH Terms: conditions — Peri-Implantitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Er:YAG laser-assisted debridement: Subjects who were randomly selected to receive debridement and surface detoxification of their implant surface and removal of the inflamed tissue with the aid of the laser treatment two years ago at the Graduate Periodontics Clinic at University of Michigan.
  Interventions: Other: Observation
- Standard mechanical debridement: Subjects who were randomly selected to receive debridement and surface detoxification of their implant surface and removal of the inflamed tissue with dental scalers two years ago at the Graduate Periodontics Clinic at University of Michigan.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Soft tissue implant measurements and radiographs

SUMMARY:
The present study represents an extension of the previously concluded randomized clinical trial "Laser-Assisted Regenerative Surgical Therapy for Peri-implantitis" (HUM00124386). The aim of the study is to compare the adjunctive effect of laser over mechanical debridement alone in the maintenance of peri-implant tissues after surgical treatment of peri-implantitis (gum disease around implants).

DETAILED DESCRIPTION:
The same 24 subjects, previously treated with surgical regenerative treatment of peri-implantitis following the LARST protocol, will be invited to return for three follow-up visits. During the follow-up visits, clinical measurements, x-rays, and pictures of the inside of their mouth will be taken to evaluate the success of their peri-implantitis treatment. If needed, additional laser treatment of the dental implant may also be provided according to the same randomization of subjects in the original study. No placebo laser application will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously enrolled subjects in the randomized clinical trial of laser-assisted regenerative surgical therapy

Exclusion Criteria:

* Unable to reach the subject
* The implant is mobile or lost

Premature Exclusion Criteria:

* The researcher believes that it is not the best interest of the subject to stay in the study
* If the subject becomes ineligible to participate based on the exclusion criteria
* If the subject's medical condition requires interventions which preclude involvement in the study (radiation therapy, chemotherapy, etc.)
* If the subject does not follow study related instructions
* The study is suspended or canceled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who previously participated in the Laser-Assisted Regenerative Surgical Therapy for Peri-implantitis study HUM00124386.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Change in Periodontal Probing Depths (PD) | Baseline and 6 months
  PD will be measured in millimeters. Change in PD measurements were calculated between baseline and 24 weeks

SECONDARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline and 6 months
  CAL will be measured in millimeters. Change in subject CAL measurements were calculated between baseline and 6 months.
Change in marginal bone level (MBL) | Baseline and 6 months
  Marginal bone level will be measured compared to baseline. Participants' standardized radiographs will be used to determine bone level changes between baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Wei Wang, DDS, DMSc, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Hashedi AA, Laurenti M, Benhamou V, Tamimi F. Decontamination of titanium implants using physical methods. Clin Oral Implants Res. 2017 Aug;28(8):1013-1021. doi: 10.1111/clr.12914. Epub 2016 Jul 8. PMID 27392811
- [Background] Albouy JP, Abrahamsson I, Persson LG, Berglundh T. Spontaneous progression of ligatured induced peri-implantitis at implants with different surface characteristics. An experimental study in dogs II: histological observations. Clin Oral Implants Res. 2009 Apr;20(4):366-71. doi: 10.1111/j.1600-0501.2008.01645.x. PMID 19309770
- [Background] Berglundh T, Wennstrom JL, Lindhe J. Long-term outcome of surgical treatment of peri-implantitis. A 2-11-year retrospective study. Clin Oral Implants Res. 2018 Apr;29(4):404-410. doi: 10.1111/clr.13138. Epub 2018 Mar 25. PMID 29575025
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Loup PJ, Heitz F, Kruger E, Lang NP. Supportive peri-implant therapy following anti-infective surgical peri-implantitis treatment: 5-year survival and success. Clin Oral Implants Res. 2018 Jan;29(1):1-6. doi: 10.1111/clr.12910. Epub 2016 Jun 23. PMID 27335316
- [Background] Isehed C, Svenson B, Lundberg P, Holmlund A. Surgical treatment of peri-implantitis using enamel matrix derivative, an RCT: 3- and 5-year follow-up. J Clin Periodontol. 2018 Jun;45(6):744-753. doi: 10.1111/jcpe.12894. Epub 2018 Apr 26. PMID 29574866
- [Background] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954
- [Background] Lin GH, Suarez Lopez Del Amo F, Wang HL. Laser therapy for treatment of peri-implant mucositis and peri-implantitis: An American Academy of Periodontology best evidence review. J Periodontol. 2018 Jul;89(7):766-782. doi: 10.1902/jop.2017.160483. PMID 30133748
- [Background] Mizutani K, Aoki A, Coluzzi D, Yukna R, Wang CY, Pavlic V, Izumi Y. Lasers in minimally invasive periodontal and peri-implant therapy. Periodontol 2000. 2016 Jun;71(1):185-212. doi: 10.1111/prd.12123. PMID 27045437
- [Background] Renvert S, Lindahl C, Persson GR. Occurrence of cases with peri-implant mucositis or peri-implantitis in a 21-26 years follow-up study. J Clin Periodontol. 2018 Feb;45(2):233-240. doi: 10.1111/jcpe.12822. Epub 2017 Nov 29. PMID 28963776
- [Background] Roccuzzo M, Layton DM, Roccuzzo A, Heitz-Mayfield LJ. Clinical outcomes of peri-implantitis treatment and supportive care: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:331-350. doi: 10.1111/clr.13287. PMID 30328195
- [Background] Roccuzzo M, Pittoni D, Roccuzzo A, Charrier L, Dalmasso P. Surgical treatment of peri-implantitis intrabony lesions by means of deproteinized bovine bone mineral with 10% collagen: 7-year-results. Clin Oral Implants Res. 2017 Dec;28(12):1577-1583. doi: 10.1111/clr.13028. Epub 2017 Jun 18. PMID 28626970
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Schwarz F, Hegewald A, John G, Sahm N, Becker J. Four-year follow-up of combined surgical therapy of advanced peri-implantitis evaluating two methods of surface decontamination. J Clin Periodontol. 2013 Oct;40(10):962-7. doi: 10.1111/jcpe.12143. Epub 2013 Aug 12. PMID 23931259
- [Background] Takagi T, Aoki A, Ichinose S, Taniguchi Y, Tachikawa N, Shinoki T, Meinzer W, Sculean A, Izumi Y. Effective removal of calcified deposits on microstructured titanium fixture surfaces of dental implants with erbium lasers. J Periodontol. 2018 Jun;89(6):680-690. doi: 10.1002/JPER.17-0389. PMID 29536538
- [Background] Wang HL, Garaicoa-Pazmino C, Collins A, Ong HS, Chudri R, Giannobile WV. Protein biomarkers and microbial profiles in peri-implantitis. Clin Oral Implants Res. 2016 Sep;27(9):1129-36. doi: 10.1111/clr.12708. Epub 2015 Oct 1. PMID 26424287